CLINICAL TRIAL: NCT07027644
Title: The Synergistic Effects of Integrated Neuromuscular Inhibition Technique and Dry Cupping Therapy on Pain Modulation and Functional Recovery on Myofascial Trigger Points of Upper Trapezius: A Randomized Controlled Trial
Brief Title: The Synergistic Effects of Integrated Neuromuscular Inhibition Technique and Dry Cupping Therapy on Pain Modulation and Functional Recovery on Myofascial Trigger Points of Upper Trapezius
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Dina Al-Amir Mohamed Hussein, Lecturer, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BeniSuefU25
Record Dates: First submitted 2025-06-11; First posted 2025-06-18 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Mechanical Neck Pain
Keywords: Dry cupping; Integrated Neuromuscular Inhibition technique

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- stretching and strengthening group (Placebo Comparator): Patients in this group will receive stretching and strengthening exercises, two sessions per week for four weeks
  Interventions: Other: stretching and strengthening exercises
- Integrated Neuromuscular Inhibition Group (Experimental): Patients in this group will receive the Integrated Neuromuscular Inhibition technique three sessions per week for four weeks
  Interventions: Other: Integrated Neuromuscular Inhibition Technique
- Dry cupping group (Experimental): Patients in this group will receive Dry cupping therapy, two sessions per week for four weeks
  Interventions: Device: Dry Cupping Therapy
- Combined treatment group (Experimental): Patients in this group will receive Dry cupping therapy, two sessions per week for four weeks, the Integrated Neuromuscular Inhibition technique, three sessions per week for four weeks plus stretching and strengthening exercises, two sessions per week for four weeks
  Interventions: Other: combined integrated neuromuscular inhibition, dry cupping and stretching and strengthening exercises

INTERVENTIONS:
Device: Dry Cupping Therapy — The patients receive dry cupping therapy for 10 min on the marked trigger point using a plastic set with a hand vacuum pump
  Arms: Dry cupping group
Other: Integrated Neuromuscular Inhibition Technique — The patients receive the Integrated Neuromuscular Inhibition Technique, which consists of ischemic compression, strain-counterstrain, and muscle energy techniques.
  Arms: Integrated Neuromuscular Inhibition Group
Other: stretching and strengthening exercises — The patients receive stretching and strengthening exercises
  Arms: stretching and strengthening group
Other: combined integrated neuromuscular inhibition, dry cupping and stretching and strengthening exercises — the patients recive all the three interventions
  Arms: Combined treatment group

SUMMARY:
The purpose of the study is to investigate the Synergistic Effects of the Integrated Neuromuscular Inhibition Technique and Dry Cupping Therapy on Pain Modulation and functional recovery on Myofascial Trigger Points of the upper trapezius

ELIGIBILITY:
Inclusion Criteria:

* Medically competent men and women will be included They had chronic MTrPs in the upper trapezius for more than 6 months Diagnostic criteria of being a tight band with a palpable nodule and distant pain when subjected to pressure

Exclusion Criteria:

* subjects with previous neck or shoulder pathology (e.g., fracture, sur¬gery, inflammatory and infectious diseases), cervical disc pathology, systemic disorder, fibromyalgia, those who underwent physical therapy for at least the previous 3 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 0-4 weeks
  pain intensity will be measured by visual analogue scale
pain pressure threshold | 0-4 weeks
  The pressure algometer will measure the pain pressure threshold

SECONDARY OUTCOMES:
Neck Disability Index | 0-4 weeks
  The Neck Disability Index is a questionnaire to measure function

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt